CLINICAL TRIAL: NCT00240149
Title: Pilot Study Evaluating Use of Insulin-Glucose Algorithm and Glucose Monitoring Techniques to Control Hyperglycemia in the Pediatric Intensive Care Unit
Brief Title: Pilot Study to Evaluate a Method of Controlling High Blood Sugar in the Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95771; Medtronic Minimed - Pending; NIH Training Grant - DK07217
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2007-12-20 (Estimated); Status verified 2007-11

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

INTERVENTIONS:
Drug: Regular Insulin via Insulin-Glucose Algorithm

SUMMARY:
Recent studies of adult intensive care unit (ICU) patients have shown significantly decreased morbidity and mortality when blood sugar concentrations are closely controlled. The safety and efficacy of this type of blood sugar management has not been studied in the pediatric ICU population. Based on the current pediatric literature data as well as our extensive retrospective study, blood sugar concentrations have a potentially profound role to play among PICU patients. In preparation for a multi-center randomized control trial, we propose a prospective feasibility study to evaluate the safety and effectiveness of using an insulin delivery algorithm to manage blood sugar in the PICU. Our hypothesis for this feasibility trial is that uniformly monitoring and controlling blood glucose with a Discrete-Closed-Loop(DCL) insulin delivery algorithm will be an effective, safe, and consistent means of delivering insulin to manage glucose in the pediatric intensive care unit.

DETAILED DESCRIPTION:
The Diabetes Control and Complications Trial (DCCT) demonstrated that long-term microvascular complications from hyperglycemia could be reduced in adolescents and adults by intensive diabetes management.1 Hyperglycemia has also been shown to be an acute risk factor for poor outcome in a variety of adult cases including trauma, cardiac,2 surgical, stroke, and head injury patients.

Moreover, control of hyperglycemia improves the outcome of these critically ill adult patients in intensive care unit (ICU) settings. In a prospective randomized study, Van den Berghe et al. reported on 1,548 patients admitted to an adult surgical ICU. During admission, intensive treatment with intravenous insulin to control hyperglycemia in both diabetics and non-diabetics reduced the risk of death by 42%, overall in-hospital mortality by 34%, sepsis by 46%, and acute renal failure by 41%.3 Utilizing less stringent criteria for glycemic control, Finney et al. also reported similar findings.4

While these studies have emphasized the value of controlling hyperglycemia in the adult ICU, there have been relatively few studies evaluating the incidence of hyperglycemia, and its correlates, in the PICU, and no interventional studies. 5,6

Because of the limited pediatric data available and the impressive findings displayed in the adult literature, we performed a retrospective chart review of all pediatric patients admitted to our PICU over a 13 month period. The goals of this study were to gain a better understanding of current glucose monitoring techniques in the PICU as well how hyperglycemia correlates with morbidity and mortality in pediatrics.

The results confirmed our hypothesis that a higher peak glucose during an admission is associated with longer LOS and a higher mortality rate. 7

As demonstrated in adults, control of hyperglycemia has the potential to have a profound impact on the morbidity and mortality of patients in the PICU. Our preliminary study clearly showed that hyperglycemia is associated with increased LOS and mortality. Unfortunately, the true clinical impact of controlling hyperglycemia on pediatric ICU patients is not known. By more accurately and more safely controlling hyperglycemia in the PICU, we have the opportunity to improve on the standard of care as well as to potentially improve the overall clinical outcome of PICU patients. Once the use of an insulin delivery algorithm and our methods for glucose monitoring have been explored in this randomized controlled feasibility study, this form of improved glucose management can be formally tested in a large multi-center trial in the PICU setting.

ELIGIBILITY:
Inclusion Criteria::

Patients between 1-18 years of age admitted to the PICU at LPCH will be asked to participate in a randomized feasibility trial during their hospitalization. This initial age restriction will be adjusted as experience is gained.

Patient displays evidence of hyperglycemia (>150mg/dl) Exclusion Criteria:Initially, patients younger than 5 years of age will be excluded. These patients appear to have a higher sensitivity to insulin as well as a proposed higher risk of hypoglycemia. Since this is a feasibility trial using insulin to control glucose, we feel that it would be prudent to establish success in an older patient population before extending the study to include younger children and infants. In addition, our PICU study revealed no significant increased risk of hyperglycemia based on age. This age restriction will be adjusted after the mid-study data analysis.

Patients who are known to be pregnant will be excluded.

Patients who have known platelet dysfunction will be excluded.

Patients without intact, uninfected skin at the future site of sensor insertion.

Study patients re-admitted to the PICU after hospital discharge will not be eligible for repeat participation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0
Dates: Start 2005-10; Study Completion 2006-03

PRIMARY OUTCOMES:
Specific Aim #1 Intervention): Randomized study of strict glucose control in a pediatric intensive care unit (PICU) using a discrete-closed-loop (DCL) insulin algorithm.
Safely reach and maintain a glucose range goal of 90-120 mg/dl in the treatment group within 4 hrs of initiating therapy.
Maintain at least 90% of glucose values within the target range.
Have fewer than 1% of glucose values below 50 mg/dl.
d) Show a significant difference in glucose values (mean glucose values and area under the curve) between the Treatment and Control group.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Buckingham, Sub-Investigator — Stanford University; Darrell M Wilson, Sub-Investigator — Stanford University
Locations (2):
- United States (2):
  - Lucile Packard Childrens Hospital - PICU, Stanford, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Finney SJ, Zekveld C, Elia A, Evans TW. Glucose control and mortality in critically ill patients. JAMA. 2003 Oct 15;290(15):2041-7. doi: 10.1001/jama.290.15.2041. PMID 14559958
- [Background] Capes SE, Hunt D, Malmberg K, Gerstein HC. Stress hyperglycaemia and increased risk of death after myocardial infarction in patients with and without diabetes: a systematic overview. Lancet. 2000 Mar 4;355(9206):773-8. doi: 10.1016/S0140-6736(99)08415-9. PMID 10711923
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Cochran A, Scaife ER, Hansen KW, Downey EC. Hyperglycemia and outcomes from pediatric traumatic brain injury. J Trauma. 2003 Dec;55(6):1035-8. doi: 10.1097/01.TA.0000031175.96507.48. PMID 14676647
- [Background] Srinivasan V, Spinella PC, Drott HR, Roth CL, Helfaer MA, Nadkarni V. Association of timing, duration, and intensity of hyperglycemia with intensive care unit mortality in critically ill children. Pediatr Crit Care Med. 2004 Jul;5(4):329-36. doi: 10.1097/01.pcc.0000128607.68261.7c. PMID 15215001
- [Background] Wintergerst KA, Deiss D, Buckingham B, Cantwell M, Kache S, Agarwal S, Wilson DM, Steil G. Glucose control in pediatric intensive care unit patients using an insulin-glucose algorithm. Diabetes Technol Ther. 2007 Jun;9(3):211-22. doi: 10.1089/dia.2006.0031. PMID 17561791